CLINICAL TRIAL: NCT02214901
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Study to Evaluate Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses BIBW 2948 BS (0.75 to 150 mg Inhalation Powder, Hard Capsule for HandiHaler®) in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of BIBW 2948 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1219.1
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Inhalation

ARMS (2):
- BIBW 2948 BS in single rising doses (Experimental)
  Interventions: Drug: BIBW 2948 BS for oral inhalation
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBW 2948 BS for oral inhalation
  Arms: BIBW 2948 BS in single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability, and pharmacokinetics of BIBW 2948 BS

ELIGIBILITY:
Inclusion Criteria:

* Healthy males based on a complete medical history, including physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests:

  * No finding deviating from normal and of clinical relevance
  * No evidence of a clinically relevant concomitant disease
* Aged between ≥21 and ≤50 years
* BMI (Body Mass Index) between ≥18.5 and ≤30 kg/m2
* Provision of written informed consent signed and dated prior to admission to the study in accordance with good clinical practice (GCP) and local legislation

Exclusion Criteria:

* Any finding during the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2005-03; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in vital signs (blood pressure, pulse rate, respiratory rate, orthostasis test, oral body temperature) | Up to 8 days after start of treatment
Changes from baseline in clinical laboratory tests | Up to 8 days after start of treatment
Changes from baseline in 12-lead electrocardiogram (ECG) | Up to 8 days after start of treatment
Number of patients with adverse events | Up to day 29
Changes from baseline in airway resistance (Raw) | Pre-dose, up to 24 hours after start of treatment
  measured via plethysmography
Assessment of tolerability by investigator, a 4-point scale | Up to 8 days after start of treatment

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analytes in plasma at different time points (AUCt1-t2) | Pre-dose, up to 48 hours after start of treatment
Maximum concentration of BIBW 3056 ZW in plasma (Cmax) | Pre-dose, up to 48 hours after start of treatment
Time from dosing to maximum concentration of the analytes in plasma (tmax) | Pre-dose, up to 48 hours after start of treatment
Amount of BIBW 3056 ZW eliminated in urine at different time points (Aet1-t2) | Pre-dose, up to 48 hours after start of treatment
Fraction of BIBW 3065 ZW eliminated in urine at different time points (fet1-t2) | Pre-dose, up to 48 hours after start of treatment
Renal clearance of BIBW 3056 ZW from 0 to 24 hours (CLR,0-24) | Pre-dose, up to 48 hours after start of treatment
Terminal rate constant of BIBW 3056 ZW in plasma (λz) | Pre-dose, up to 48 hours after start of treatment
Terminal half life of BIBW 3056 ZW in plasma (t½) | Pre-dose, up to 48 hours after start of treatment
Mean residence time of BIBW 3056 ZW in the body after inhalation (MRTih) | Pre-dose, up to 48 hours after start of treatment
Apparent clearance of BIBW 3056 ZW in the plasma after extravascular administration (CL/F) | Pre-dose, up to 48 hours after start of treatment
Apparent volume of distribution of BIBW 3056 ZW during the terminal phase λz following an extravascular dose (Vz/F) | Pre-dose, up to 48 hours after start of treatment
The percentage of the AUC 0-∞ that is obtained by extrapolation (%AUCtz-∞) | Pre-dose, up to 48 hours after start of treatment